CLINICAL TRIAL: NCT01362400
Title: A Phase 2, Double-Blind, Placebo-Controlled Study of IPI-504 and Docetaxel in Previously Treated Patients With Stage IIIB or IV Non-Small Cell Lung Cancer
Brief Title: A Double-blind Study Evaluating IPI-504 and Docetaxel in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPI 504-14
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: LUNG NEOPLASMS; LARGE CELL CARCINOMA; SQUAMOUS CELL CARCINOMA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Carcinoma, Large Cell; Carcinoma, Squamous Cell | interventions — tanespimycin; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM 1: IPI 504 + Docetaxel (Active Comparator): Drug: IPI-504 plus Docetaxel
  Interventions: Drug: IPI 504 plus Docetaxel
- Placebo + Docetaxel (Placebo Comparator): Placebo plus Docetaxel
  Interventions: Drug: Placebo plus Docetaxel

INTERVENTIONS:
Drug: IPI 504 plus Docetaxel — 450 mg/m2 (starting dose) IPI-504 or placebo IV (in the vein) day 1, 8 & 15 during each 21 day cycle
  75 mg/m2 in US and EU, 60 mg/m2 in South Korea and Taiwan Docetaxel (Taxotere®) will be administered by IV infusion every 3 weeks (Day 1 of each 21-day cycle)
  Other Names: IPI-504; Docetaxel
  Arms: ARM 1: IPI 504 + Docetaxel
Drug: Placebo plus Docetaxel — 450 mg/m2 (starting dose) IPI-504 or placebo IV (in the vein) day 1, 8 & 15 during each 21 day cycle
  75 mg/m2 in US and EU, 60 mg/m2 in South Korea and Taiwan Docetaxel (Taxotere®) will be administered by IV infusion every 3 weeks (Day 1 of each 21-day cycle)
  Other Names: Docetaxel
  Arms: Placebo + Docetaxel

SUMMARY:
The purpose of this study is to compare the impact of IPI-504 in combination with docetaxel to placebo in combination with docetaxel on life expectancy in patients with Non Small Cell Lung cancer (NSCLC). Docetaxel is an approved chemotherapy for NSCLC. An additional goal of the study is to determine the effect of IPI-504, in combination with docetaxel, verses placebo in, combination with docetaxel, on the growth of cancer

DETAILED DESCRIPTION:
This is a Phase 2, double-blind, randomized, placebo-controlled study in patients with previously treated, locally advanced or metastatic Stage IIIb or IV NSCLC designed to compare IPI-504 plus docetaxel versus placebo plus docetaxel. All patients will have at least a 15 pack year smoking history. Tumor samples will be assessed by a central pathology reviewer to confirm pathology that is documented at baseline; this review need not occur in advance of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years of age
* Voluntarily signed an informed consent
* Confirmed NSCLC and Stage IIIB or IV disease.
* At least a ≥15 pack year smoking history and must have been an active smoker within 20 years of diagnosis.
* Must have archival NSCLC tissue available to provide for analysis or have a lesion that is accessible for biopsy
* Must have experienced disease progression during or after receiving at least 1 prior platinum-containing chemotherapy regimen.
* Must have received no more than 2 prior chemotherapy regimens
* Measurable disease by RECIST 1.1 criteria.
* ECOG performance status of 0 or 1 (Refer to scale in Appendix 1).
* Women of child-bearing potential (WCBP), all sexually active male patients, and partners of patients must agree to use adequate methods of birth control.

Exclusion Criteria:

* Prior docetaxel, IPI-504 or other Hsp90 inhibitor treatment
* Known hypersensitivity to drugs formulated with polysorbate-80.
* Not recovered from any toxicities related to prior treatment
* Use of a medication or food that is a clinically relevant CYP3A inhibitor or inducer
* Inadequate hematologic function
* Inadequate hepatic function
* Inadequate renal function
* Symptomatic keratitis or keratoconjunctivitis.
* Uncontrolled systemic fungal, bacterial, viral or other infection
* Patients with clinically active brain metastases
* Patients with clinically stable brain metastases (previously treated or untreated) are eligible.
* Sinus bradycardia (resting heart rate <50 bpm).
* Significant cardiac disease
* Previous or current malignancies at other sites within the last 2 years
* Prior hepatic resections or hepatic-directed therapy
* Known HIV-positive patients receiving combination antiretroviral therapy.
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2011-05; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Up to three years from last patient study visit
  To determine the overall survival rate of patients administered IPI-504 plus docetaxel vs. placebo plus docetaxel

SECONDARY OUTCOMES:
Progression Free Survival | Up to three years from last patient study visit
  To determine the progression free survival rate from randomization to progression or death whichever occurs first, of all patients and in a subpopulation of patients administered IPI-504 plus docetaxel versus placebo plus docetaxel
Overall Response Rate | Up to three years from last patient study visit
  To determine partial response or complete response occurring at any point post-treatment
Time to Progression | Up to three years from last patient study visit
  To identify the amount of time from randomization to progression, of all patients and in a subpopulation of patients administered IPI-504 plus docetaxel versus placebo plus docetaxel

CONTACTS AND LOCATIONS:
Overall Officials: Tess Schmalbach, MD, Study Director — Infinity Pharmaceuticals, Inc.
Locations (64):
- United States (41):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - University of California Irvine Medical Center, Orange, California
  - PMK Medical Group, Inc., Oxnard, California
  - Wilshire Oncology Medical Group, Inc., Rancho Cucamonga, California
  - American Institute of Research, Whittier, California
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists and Research Institute, St. Petersburg, Florida
  - Central Indiana Cancer Centers, Carmel, Indiana
  - Indiana University, Indianapolis, Indiana
  - Indiana University Health Ball Memorial Hospital, Muncie, Indiana
  - Community Hospital, Munster, Indiana
  - Floyd Memorial Cancer Center of Indiana, New Albany, Indiana
  - Owsley Brown Frazier Cancer Center-Louisville Downtown, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ann Arbor Hematology Oncology Associates, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Metro Health Cancer Center, Wyoming, Michigan
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Broome Oncology, LLC, Johnson City, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Piedmont Hematology Oncology Associates, PLLC, Winston-Salem, North Carolina
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Cancer Centers of the Carolinas, Seneca, South Carolina
  - Chattanooga Oncology and Hematology Associates, PC, Chattanooga, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Texas Oncology-Arlington South, Arlington, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - Virginia Cancer Institute, Richmond, Virginia
  - Puget Sound Cancer Centers, Edmonds, Washington
- Hungary (5):
  - Pándy Kálmán Megyei Kórház, Gyula, Bekes County
  - Sopron MJV Erzsébet Kórház, A DEOEC Oktató Kórháza, Sopron, Győr-Moson-Sopron
  - Mátrai Gyógyintézet, Mátraháza, Heves County
  - Zala Megyei Kórház, Zalaegerszeg, Zala County
  - Országos Korányi TBC és Pulmonológiai Intézet, Budapest
- Romania (4):
  - Institutul Oncologic "Prof. Dr. I. Chiricuta", Cluj-Napoca, Cluj
  - Spitalul de Urgenta "Constantin Opris", Baia Mare, Maramureş
  - Spitalul Municipal Ploiesti, Ploieşti, Prahova
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu, Sibiu County
- Russia (4):
  - City Oncology Hospital # 62, Moscow Region, Moscow
  - State Budget Institution of Healthcare "Chelyabinsk Regional Clinical Oncology Dispensary", Chelaybinsk
  - Blokhin Cancer Research Center of Russia, Dept. of clinical pharmacology, Moscow
  - Non-State Central Clinical Hospital # 2 named N.A. Semashko of "OAO RGD", Moscow
- South Korea (6):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Inha University Hospital, Jung Gu, Incheon
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Dong-A University Medical Center, Busan
  - Severance Hospital,Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei